CLINICAL TRIAL: NCT05174962
Title: National Stigma Survey About Mental Illness, Homelessness and Intellectual Disability in Spain
Brief Title: National Stigma Survey About Mental Illness, Intellectual Disability and Homelessness in Spain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Grupo 5 (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020/21-026
Record Dates: First submitted 2021-11-17; First posted 2022-01-03 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-10

CONDITIONS: General Population
Keywords: Stigma; Mental illness; Homeless situation; Intellectual disability
MeSH Terms: conditions — Social Stigma; Mental Disorders; Intellectual Disability

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project is framed within the "Complutense University of Madrid (UCM)-Group 5 Against Stigma Chair", of the Faculty of Psychology. The main objective of the Chair is to fight the stigma that affects people with mental disorders, disabilities, vulnerability or extreme social exclusion. For this purpose, the Chair is developing research studies, training programs, cultural activities and awareness campaigns, proof of this is the recent publication of the Guide to good practices against stigma, which, although it takes as a reference to the people with a diagnosis of mental disorder, it is expected to be generalizable to other groups.

Stigma is associated with the condition of being different, and affects any person belonging to a minority or vulnerable group, being one of the main obstacles to full participation in different social, political and cultural institutions. The fight against stigma is included in important international treaties, such as the United Nations Convention on the Rights of Persons with Disabilities or the European recommendations regarding the fight against social exclusion of people with mental health problems.

This study will focus on three groups of special social sensitivity, with clear stigmatizing conditions: people with mental health problems, people in a homeless situation and people with intellectual disabilities.

DETAILED DESCRIPTION:
The primary aim of this research is to describe the stigma faced by people corresponding to three highly vulnerable population groups: people with mental health problems, homeless people and people with intellectual disabilities.

From this general aim, four different specific goals are derived: 1) To delve into the experience of stigma of these groups, from first person; 2) To develop a quantitative assessment instrument that captures the current needs and experiences of people from these groups; 3) To describe and compare the social stigma of these three groups in a representative Spanish sample; 4) To address, from a gender perspective, possible differences in terms of the variables explored in the populations under study.

ELIGIBILITY:
Inclusion Criteria:

* People aged 18 and over from general population.
* Any gender.

Exclusion Criteria:

* People under 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: An approximate sample size of 2750 interviews is estimated. The sample made up of the general population over 18 years of age obtained through the consumer panel methodology.
  To obtain a representative sample of the Spanish population, quotas by sex and age group are included, as well as data for each of the 17 autonomous communities through simple affixing, ensuring a minimum of 100 surveys per Autonomous Community. On the other hand, it also allows a rural-urban analysis in the sample as a whole and in the most populated autonomous communities.
Sampling Method: Probability Sample
Enrollment: 2750 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Social distance desire | Up to 8 weeks
  Reported and Intended Behaviour Scale (RIBS). The scale was adapted by asking about future intentions to live with, have friendships with or let children interact with people with mental health problems, homelessness or intellectual disabilities. Responses consisted of Likert-type items (1 strongly agree, 5 strongly disagree). Higher scores are indicative of better future behaviour.
Attitudes towards mental disorders | Up to 8 weeks
  Attributional Questionnaire-9 (AQ-9). It is a reduced version of the Attribution Questionnaire-27, consisting of 9 items instead of 27. The questionnaire includes 9 items in Likert-type format with 9 response alternatives ranging from "1 = not at all" to "9 = very much".
Attitudes towards disability | Up to 8 weeks
  Attitudes to Disability Scale (ADS): This scale is one of the most complete scales for assessing stigma towards intellectual disability. It was developed as part of an international World Health Organization study, in which Spain participated alongside other countries. The scale consists of 16 Likert-type items (1 = strongly agree and 5 = strongly disagree). These items are gathered in 4 subscales: Inclusion-exclusion, Discrimination, Gains and Hopes. It has adequate psychometric properties.
Attitudes towards homelessness | Up to 8 weeks
  Survey attitudes towards Homeless People: This scale consists of 9 Likert-type items (1 = strongly agree and 6 = strongly disagree). It explores various attitudes towards homeless people (people sleeping on the streets or in shelters). It has good psychometric properties.
Disclosure about mental disorders | Up to 8 weeks
  This scale assess opinions and attitudes towards disclosure of mental health problems, as well as the ability to talk about them and to identify the main agents and sources of support for people, through this question: "If a close person (family member, friend, partner) had a mental health problem...? ". Questions are rated on a 5 Likert-type scale, where 1 = I would definitely talk about it with them, and 5 = I would avoid talking about it with them.
Key aspects of stigma | Up to 8 weeks
  In addition to the standardized instruments, a number of selected questions on key aspects of stigma are included in the survey. These qualitative aspects were highlighted by people with mental illness, people experiencing homelessness, and people with intellectual disabilities who participated in a series of focus groups. Questions are rated on a 5 Likert-type scale (1 = strongly disagree and 5 = strongly agree)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Muñoz, Ph.D., Study Chair — Universidad Complutense de Madrid; Manuel Muñoz, Ph.D., Principal Investigator — Universidad Complutense de Madrid

IPD SHARING:
Plan to Share IPD: Undecided